CLINICAL TRIAL: NCT01412710
Title: The Effect of Vitamin D Supplementation on Cardiovascular Risk Factors Among Hispanics and African Americans With Type 2 Diabetes
Brief Title: Vitamin D Supplementation on Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Principal Investigator, Fatma Ercanli-Huffman, Dr. Fatma G. Huffman, Florida International University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIU-032511-01
Record Dates: First submitted 2011-08-07; First posted 2011-08-09 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Cholecalciferol; Vitamin D; Insulin resistance; Cardiovascular disease risk; Minorities
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4000 IU group (Experimental): This group will be given 4000 IU of vitamin D3 once daily, orally for 6 months.
  Interventions: Drug: Cholecalciferol
- 6000 IU group (Experimental): This group will be given 6000 IU vitamin D3 once daily, orally for 6 months.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — 4000 IU or 6000 IU given vitamin D3 once daily, orally for 6 months.
  Other Names: Vitamin D

SUMMARY:
The purpose of the present pilot study is to determine the effect of vitamin D supplementation (4000 IU or 6000 IU once daily for 6 months) on reducing heart disease risk and in improving blood glucose control in type 2 Diabetes subjects . The investigators are working with Hispanics and African Americans living in Miami, Florida.

DETAILED DESCRIPTION:
Insufficient vitamin D levels have been found in subjects with type 2 diabetes (T2D). Similarly, a negative association between serum vitamin D levels and insulin resistance has been reported in a large sample representative of the adult US population and in subjects at risk for T2D. In addition, a strong association between hypovitaminosis D and hypertriglyceridemia has been demonstrated in studies done in US adult population.

Literature has indicated that subjects with T2D and insulin resistance (IR) are more likely to develop arteriosclerosis and all of the complications related to this condition, such as myocardial infarction and stroke.

These findings have increased the interest about the effect of vitamin D on metabolic abnormalities grouped under the term "cardiovascular disease (CVD) risk factors", which includes hypertension, dyslipidemia, obesity, glucose intolerance, inflammation and T2D which is in itself a risk factor for CVD.

Therefore, the purpose of the present pilot study will be to determine the effect of supplemental vitamin D intake (4000 IU or 6000 IU of Cholecalciferol daily for 6 months) on CVD risk markers and glycemic control; primarily lipid panel, insulin resistance, and glycosylated hemoglobin (A1C), in a sample of Hispanics and African-Americans with T2D and vitamin D insufficiency. If repletion of vitamin D level improves insulin resistance, glycemic control, inflammation, hypertension, dyslipidaemia or kidney functions, it may prevent the development of CVD events and decrease T2D complications.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* African American or Hispanic
* able to ambulate on their own
* aged between 30 - 70 years

Exclusion Criteria:

* Taking Supplemental Vitamin D
* Pregnant or Lactating women
* Receiving insulin therapy
* Not participating in other drug trials
* HIV/ hepatitis/ cancer/ liver disease/ heart failure/ any recent surgery/ mental illness/ epilepsy/ any GI or malabsorption disorders
* Kidney failure or on dialysis

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fatma G Huffman, PhD, Principal Investigator — Florida International University
Locations (1):
- Human Nutrition Laboratory, Florida International University, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from two clinics in Miami-Dade County, Florida (Borinquen Health Care Center and Clinical Care Medical Center) from July 2011 to March 2013 using flyers explaining the purpose of the study.
Pre-assignment Details: 15 participants did not qualified due to normal levels of serum vitamin D, 25-hydroxy vitamin D [25(OH)D].
Groups:
- 4000 IU Group: This group received 4000 IU/day vitamin D3 for 6 months.
- 6000 IU Group: This group received 6000 IU/day vitamin D3 for 6 months.
Period: Overall Study
Arm/Group | 4000 IU Group | 6000 IU Group
Started | 50 | 27
Completed | 46 | 22
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Population: Hispanic or Latino and African-Americans, age 30-70 years old, with type 2 diabetes.
Groups:
- 4000 IU Group: This group will be given cholecalciferol 4000 IU once daily, orally for 6 months.
- 6000 IU Group: This group will be given cholecalciferol 6000 IU once daily, orally for 6 months.
- Total: Total of all reporting groups
Arm/Group | 4000 IU Group | 6000 IU Group | Total
Number analyzed (Participants) | 50 | 27 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 23 | 67
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.76 (8.56) | 54.17 (10.99) | 54.46 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 15 | 50
  Male | 15 | 12 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 25 | 65
  Not Hispanic or Latino | 10 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 27 | 77

OUTCOME MEASURES:

1. Primary Outcome: Blood Lipid
Description: Total cholesterol will be used as surrogate measures for cardiovascular disease risk.
Time Frame: Baseline
Population: Total cholesterol baseline.
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- 4000 IU Group: Vitamin D 4000 IU/day
- 6000 IU Group: Vitamin D 6000 IU/day
Arm/Group | 4000 IU Group | 6000 IU Group
Number analyzed (Participants) | 50 | 27
mg/dl | 213.08 (42.30) | 193.88 (41.03)

2. Secondary Outcome: Glycemic Control
Description: hemoglobin A1C blood test
Time Frame: Baseline
Population: A1C baseline.
Measure: Mean (Standard Deviation); unit: Percentage of Hemoglobin
Arm/Group | 4000 IU Group | 6000 IU Group
Number analyzed (Participants) | 50 | 27
Percentage of Hemoglobin | 8.25 (2.40) | 8.26 (1.92)

ADVERSE EVENTS:
Time Frame: Data were collected for 6 months
Description: No adverse events or signs of toxicity reported by any of the participants throughout the study.
Groups:
- 4000 IU Vitamin D3/Day: This group will be given cholecalciferol 4000 IU once daily, orally for 6 months.
- 6000 IU Vitamin D3/Day: This group will be given cholecalciferol 6000 IU once daily, orally for 6 months.
Arm/Group | 4000 IU Vitamin D3/Day | 6000 IU Vitamin D3/Day
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/27
Other Adverse Events (participants affected / at risk) | 0/50 | 0/27

LIMITATIONS AND CAVEATS:
The study sample was a convenience sample and was not randomly selected from the general adult population. The study lacked a control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes